CLINICAL TRIAL: NCT04114461
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover Study to Evaluate the Safety and Pharmacokinetics of HL-TOF Tab. 5 mg Compared With Those of XelJanz Tab. in Healthy Volunteers
Brief Title: Study to Evaluate HL-TOF Tab. 5 mg Compared With XelJanz Tab. in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HL-TOF-101
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: 2X2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HL-TOF tab. 5mg (Experimental): Tofacitinib freebase
  Interventions: Drug: HL-TOF tab. 5mg
- Xeljanz tab. 5mg (Active Comparator): Tofacitinib citrate (5mg as tofacitinib)
  Interventions: Drug: Xeljanz tab. 5mg

INTERVENTIONS:
Drug: HL-TOF tab. 5mg — HL-TOF
  Other Names: Tofacitinib freebase
  Arms: HL-TOF tab. 5mg
Drug: Xeljanz tab. 5mg — Xeljanz
  Other Names: Tofacitinib citrate
  Arms: Xeljanz tab. 5mg

SUMMARY:
To evaluate the safety and pharmacokinetics of HL-TOF tab. 5 mg compared with those of XelJanz tab. in healthy volunteers

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and pharmacokinetics of tofacitinib after single oral administration of Xeljanz tab. 5mg as reference drug and HL-TOF tab. 5mg as test drug in healthy voluteers. AUC and Cmax would be evaluated for the pharmacokinetics. Adverse event, Laboratory examination and other examination result would be evaluated for the safety.

ELIGIBILITY:
Inclusion Criteria:

* Years 19-60
* No pathological symptoms or findings
* Suitable for the criteria for examination
* 90≤SBP≤139, 60≤DBP≤89
* Body weight≥50kg (Female≥45kg) and 18≤BMI≤30kg/m2
* Contraceptive during the study period
* Volunteer for the study and sign to ICF

Exclusion Criteria:

* Subject with medical history which affect on the absorption of drug
* Following condition: Mental illness, Hepatic disorder, Tuberculosis, ANC< 500cells/mm3, ALC<500cells/mm3, Hb<8g/dL
* Subject with hypersensitivity reaction to HL-TOF and Xeljanz
* Subject with galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Subject who take a vaccination within 30 days
* Subject who take a medication such as barbiturates within 30 days
* Subject who take a medication that affect to the pharmacokinetics of drug within 10 days
* Subject who take alcohol more than 21 cups per week
* Subject who smoke 20 cigarettes per day
* Subject who participate in any clinical investigation within 6 month prior to study medication dosing
* Subject with whole blood donation within 60 days, component blood donation within 14 days, blood donation within 30 days
* Subject with decision of non-participation through investigator's review

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 hour, 0.17 hour, 0.34 hour, 0.5 hour, 0.67 hour, 0.83 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 9 hour, 12 hour
  Maximum concentration
AUC | 0 hour, 0.17 hour, 0.34 hour, 0.5 hour, 0.67 hour, 0.83 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 9 hour, 12 hour
  Area under curve

SECONDARY OUTCOMES:
AE | 0 hour, 0.17 hour, 0.34 hour, 0.5 hour, 0.67 hour, 0.83 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 9 hour, 12 hour
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: JAEWOO KIM, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- YANGJI Hospital, Seoul, South Korea